CLINICAL TRIAL: NCT00896857
Title: Breast Cancer Prevention by Inducing Apoptosis in DCIS Using Breast Ductal Lavage
Brief Title: Studying Cells Collected Through Ductal Lavage in Women Undergoing Surgery for Ductal Carcinoma In Situ or Other Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU-74A04; CDR0000579246 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG04-063
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: breast duct lavage

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is evaluating cells collected through ductal lavage in women undergoing surgery for ductal carcinoma in situ or other breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the expression pattern of the programmed cell death (PCD) regulatory genes bcl-2, bax, and bcl-xL in primary ductal carcinoma in situ (DCIS) cultures.
* Determine whether down-regulation by genetic manipulation of the anti-apoptotic genes bcl-2 and/or bcl-xL, alone or in conjunction with physiological preventive doses of tamoxifen citrate, has the highest induction of PCD in primary DCIS cell cultures.
* Determine the expression pattern of the PCD regulatory genes bcl-2, bax, and bcl-xL in cells obtained by breast ductal lavage.
* Determine whether down-regulation by genetic manipulation of the anti-apoptotic genes bcl-2 and/or bcl-xL, alone or in conjunction with physiological preventive doses of tamoxifen citrate, has the highest induction of PCD in cells obtained by breast ductal lavage.

OUTLINE: Patients undergo breast lavage to collect primary epithelial cells for cytological analysis before a planned surgical procedure. Ductal carcinoma in situ (DCIS) tissue samples obtained from surgery are used to establish primary DCIS cell cultures. The DCIS cells and primary epithelial cells obtained by ductal lavage are analyzed for endogenous protein levels of bcl-2, bax, and bcl-xL, using western blotting and immunohistochemical staining, to determine the appropriate antisense oligonucleotide molecule that will be used to induce apoptosis. The DCIS cells and primary epithelial cells obtained by ductal lavage are treated with antisense oligonucleotides and/or a physiological chemopreventive dose of tamoxifen citrate to determine which will provide the highest induction of cell death. The effect of these treatments on protein expression is analyzed by western blotting and immunohistochemistry. The effect of these treatments on markers of programed cell death (PCD) (i.e., DNA fragmentation and caspase activation) is also analyzed. Changes in mRNA expression are analyzed using a PCR-based quantitation assay.

Results from the molecular marker assays are not provided to the patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Agrees to undergo breast surgical procedure AND meets one of the following criteria:

  * Scheduled to undergo breast biopsy based on suspicious mammographic or clinical breast examination findings
  * Diagnosis of ductal carcinoma in situ (DCIS) or carcinoma in the breast to be studied (opposite breast may also be studied)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Pre- or post-menopausal
* Not currently pregnant or pregnant within the past 12 months
* Must not have lactated within the past 12 months
* No active infection or inflammation in the breast to be studied
* No known allergy to lidocaine, prilocaine, or marcaine (bupivacaine)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior subareolar surgery or other breast procedure that may disrupt the ductal system within 2 cm of the nipple in the breast to be studied
* No prior breast implant that disrupts the ductal architecture in the breast to be studied
* No prior silicone injections in the breast to be studied
* No prior radiotherapy to the breast to be studied
* No chemotherapy within the past 6 months

  * Concurrent prophylactic chemotherapy allowed
* No concurrent participation in another research study that may conflict with or affect the outcome of this study

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women Undergoing Surgery for Ductal Carcinoma In Situ or Other Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Expression pattern of the programmed cell death (PCD) regulatory genes bcl-2, bax, and bcl-xL in primary ductal carcinoma in situ (DCIS) cultures
Induction of PCD by antisense oligonucleotides and/or tamoxifen citrate in primary DCIS cell cultures
Expression pattern of the PCD regulatory genes bcl-2, bax, and bcl-xL in cells obtained by breast ductal lavage
Induction of PCD by antisense oligonucleotides and/or tamoxifen citrate in cells obtained by breast ductal lavage

CONTACTS AND LOCATIONS:
Overall Officials: Patrick P. Koty, PhD, Study Chair — Wake Forest University Health Sciences